CLINICAL TRIAL: NCT05377489
Title: A Single-arm, Open-label, Phase III Trial to Evaluate the Safety and Tolerability of Intra-articular Injections of RTX-GRT7039 in Subjects With Moderate to Severe Pain Associated With Osteoarthritis of the Knee.
Brief Title: Open-label Trial to Check the Safety and Tolerability of RTX-GRT7039 Injections for Pain Associated With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF7039-03; 2021-005046-15 (EudraCT Number); U1111-1268-7230 (Other: Universal Trial Number); 2024-515709-24-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis
Keywords: Knee; Osteoarthritis; Pain assessment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RTX-GRT7039 (Experimental): Participants will receive injections of RTX-GRT7039 into either the index knee (affected knee or in case of bilateral OA the knee with highest pain intensity), or each of both knees up to Week 52.
  Interventions: Drug: RTX-GRT7039

INTERVENTIONS:
Drug: RTX-GRT7039 — RTX-GRT7039 monoarticular injections or bilateral intra-articular injections.

SUMMARY:
An open-label, single-arm clinical trial to confirm the safety of monoarticular injections or bi-lateral intra-articular injections of RTX-GRT7039 in patients who have pain associated with osteoarthritis of the knee despite standard of care.

DETAILED DESCRIPTION:
This trial comprises a total observation period of up to 78 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has given written informed consent to participate.
* The participant is 18 years of age or older at the Screening Visit.
* The participant has a diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria and functional capacity class of I to III.
* There is a documented history indicating that participant has insufficient pain relief with previous Standard of Care.

Exclusion Criteria:

* The participant has past joint replacement surgery of the index knee.
* The participant has a history of significant trauma or surgery (e.g., open or arthroscopic) to the index knee within 12 months of Screening.
* The participant has periarticular pain at the index knee from any cause other than osteoarthritis, including referred pain, bursitis, tendonitis.
* The participant has clinical hip osteoarthritis on the side of the index knee.
* The participant has a history of osteonecrosis, subchondral insufficiency fracture, atrophic osteoarthritis, rapidly progressing osteoarthritis (RPOA) Type I or Type II,pathologic fracture, primary or metastatic tumor, or joint infection in the index knee.
* The participant has significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus >10°, valgus >10°) by radiograph as assessed by independent Central Readers at Screening Visit.
* The participant has other conditions that could affect trial endpoint assessments of the index knee.
* The participant has current clinically significant disease(s) or condition(s) that may affect safety assessments, or any other reason which may preclude the participant's participation for the full duration of the trial.
* The participant has a history of hypersensitivity to resiniferatoxin (RTX) or any similar component (capsaicin, chili peppers).
* The participant is currently participating or was participating in another investigational drug trial within 3 months prior to the Screening Visit.
* The participant is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site or is a family member of the employees or the investigator.

The non-index knee is not eligible for treatment in the trial, if any of the knee-related exclusion criteria applies to the non-index knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (27):
  - Arizona Arthritis and Rheumatology Associates (AARA) P.C, Glendale, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Orange County Research Institute, Anaheim, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - Westlake Medical Research, Thousand Oaks, California
  - Progressive Medical Research, Port Orange, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - OrthoIndy, Inc., Greenwood, Indiana
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Oakland Medical Research Center, Troy, Michigan
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - M3-Emerging Medical Research, LLC, Raleigh, North Carolina
  - University Orthopedics Center, State College, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Accellacare-Knoxville, Knoxville, Tennessee
  - Tekton Research, Inc., San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
- Bulgaria (10):
  - UMHAT Eurohospital Plovdiv OOD, Plovdiv
  - Medical Centre Artmed, Plovdiv
  - MHAT Kaspela EOOD, Plovdiv
  - UMHAT Pulmed, Plovdiv
  - University Multiprofile Hospital For Active Treatment Pulmed OOD, Plovdiv
  - Medical Centre N. I. Pirogov EOOD, Sofia
  - MHAT St Iv. Rilski, Sofia
  - UMBAL Sveti Ivan Rilski EAD, Sofia
  - Synexus Medical Center Sofia, Sofia
  - Multi-Profile District Hospital for Active Treatment Dr. Stefan Cherkezov, Veliko Tarnovo
- Japan (6):
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Medical Corporation Kouhoukai Takagi Hospital, Okawa-shi, Fukuoka
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Saiseikai Kanagawaken Hospital, Yokohama, Kanagawa
  - Otakibashi Orthopedic Clinic, Shinjuku-ku, Tokyo
  - Saitama Medical Center, Saitama
- Poland (21):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne 4M Plus, Krakow, Malopolska
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - ClinicMed Badurski I Wspolnicy Spolka Jawna, Bialystok
  - ClinicMed Daniluk, Nowak Spolka komandytowa, Bialystok
  - Zaklad Opieki Zdrowotnej w Boleslawcu, Bolesławiec
  - Centrum Kliniczno, Elblag
  - NZOZ Medi Spatz, Gliwice
  - PZU Zdrowie S.A. Oddzia¿ Centrum Medyczne Artimed w Kielcach, Kielce
  - Centrum Medyczne Semper fortis, Krakow
  - Centermed Krakow Sp. z o.o., Krakow
  - Nzoz Centermed Krakow, Szpital I Przychodnia, Krakow
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Medyczne Centrum Hetmanska Indywidualna Specjalistyczna Praktyka Lekarska Dr Hab Piotr Leszczynski, Poznan
  - Medyczne Centrum Hetmanska, Poznan
  - RCMed Oddzial Sochaczew, Sochaczew
  - RCMed Piotr Opadczuk, Sochaczew
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - ETG Warszawa, Warsaw
  - Europejskie Centrum leczenia Chorob Cywilizacyjnych, Warsaw
  - Wojewodzki Szpital Zespolony W Kielcach, Kielce, Świętokrzyskie Voivodeship
- Romania (9):
  - Spitalul Judetean Caracal, Caracal, Olt
  - SC Medicali's SRL, Timișoara, Timiș County
  - SC Medaudio-Optica SRL, Râmnicu Vâlcea, Vâlcea County
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - SC Centrul Medical Sana SRL, Bucharest
  - Spitalul Clinic Sf. Maria, Bucharest
  - Spital Clinic Dr I Cantacuzino, Bucharest
  - SC Policlinica CCBR SRL, Bucharest
  - Sf. Maria Hospital, Bucharest
- South Africa (18):
  - Tread Research, Parow, Cape Town
  - Tygerberg hospital, Parow, Cape Town
  - Josha Research, Bloemfontein, Free State
  - Welkom Clinical Trial Centre, Welkom, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Midrand Medical Centre, Halfway House, Gauteng
  - Lakeview Hospital, Johannesburg, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - University of Pretoria, Pretoria, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Sandton Medical Research (Newtown CRC), Sandton, Gauteng
  - Clinresco Centres (Pty) Ltd., Kempton Park, Johannesburg
  - Synapta Clinical Research Center, Durban, KwaZulu-Natal
  - Dr Zubar Fazal Ahmed Vawda MD, Durban, KwaZulu-Natal
  - Precise Clinical Solutions, Durban, KwaZulu-Natal
  - Aliwal Shoal Medical Centre, eMkhomazi, KwaZulu-Natal
  - Medicross Langeberg Medical & Dental Centre, Kraaifontein, Western Cape
  - Arthritis Clinical Research Centre, Cape Town
- United Kingdom (3):
  - Accellacare Yorkshire, Shipley, Yorkshire
  - Accellacare Warwickshire, Coventry
  - Chapel Allerton Hospital - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
URL: https://www.grunenthal.com/en/science/clinical-trials/data-sharing-clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- RTX-GRT7039: * RTX-GRT7039 was administered as an intra-articular injection or repeated intra-articular injections of RTX-GRT7039 in participants with moderate to severe pain associated with osteoarthritis (OA) of the knee, despite receiving continued treatment with optimal standard-of-care (SoC) or who are unable to receive SoC treatment due to contraindications or intolerability.
  * Participants received injections of RTX-GRT7039 into either the index knee (affected knee or in case of bilateral OA the knee with higher pain severity), or both knees up to Week 52.
  * Participants received up to four repeated injections between 3 and 12 months after the first injection based on the persistence or return of pain, with a minimum interval of 12 weeks between injections.
Period: Overall Study
Arm/Group | RTX-GRT7039
Started | 714
Completed | 539
Not Completed | 175
Not completed — Withdrawal by Subject | 122
Not completed — Lost to Follow-up | 21
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 5
Not completed — Death | 4
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Groups:
- RTX-GRT7039: * RTX-GRT7039 was administered as an intra-articular injection or repeated intra-articular injections of RTX-GRT7039 in participants with moderate to severe pain associated with OA of the knee, despite receiving continued treatment with optimal SoC or who are unable to receive SoC treatment due to contraindications or intolerability.
  * Participants received injections of RTX-GRT7039 into either the index knee (affected knee or in case of bilateral OA the knee with higher pain severity), or both knees up to Week 52.
  * Participants received up to four repeated injections between 3 and 12 months after the first injection based on the persistence or return of pain, with a minimum interval of 12 weeks between injections.
Arm/Group | RTX-GRT7039
Number analyzed (Participants) | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 548
  Male | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 52
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 75
  White | 574
  More than one race | 10
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: From Baseline up to Week 78
Measure: Count of Participants; unit: Participants
Arm/Group | RTX-GRT7039
Number analyzed (Participants) | 714
Participants | 394

2. Primary Outcome: Number of Participants With TEAEs Leading to Study Discontinuation
Time Frame: From Baseline up to Week 78
Measure: Count of Participants; unit: Participants
Arm/Group | RTX-GRT7039
Number analyzed (Participants) | 714
Participants | 9

3. Secondary Outcome: Number of Participants With TEAEs Representing Structural Changes as Assessed by Imaging Methods
Time Frame: From Baseline up to Week 78
Measure: Count of Participants; unit: Participants
Arm/Group | RTX-GRT7039
Number analyzed (Participants) | 714
Participants | 7

4. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Score
Description: The WOMAC pain subscale will be assessed using an 11-point numerical rating scale (NRS), where 0= no pain and 10=worst pain.
Time Frame: From Baseline up to Week 12
Population: Results reported separately for Index Knee and Non-index Knee
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX-GRT7039
Number analyzed (Participants) | 698
units on a scale
  Index Knee | -2.73 (2.053)
  Non-index Knee: number analyzed (Participants) | 279
  Non-index Knee | -2.33 (1.944)

ADVERSE EVENTS:
Time Frame: Up to 78 weeks
Groups:
- RTX-GRT7039: * RTX-GRT7039 was administered as an intra-articular injection or repeated intra-articular injections of RTX-GRT7039 in participants with moderate to severe pain associated with osteoarthritis (OA) of the knee, despite receiving continued treatment with optimal standard-of-care (SoC) or who are unable to receive SoC treatment due to contraindications or intolerability.
  * Participants received injections of RTX-GRT7039 into either the index knee (affected knee or in case of bilateral OA the knee with highest pain severity), or each of both knees up to Week 52.
  * Participants received up to four repeated injections between 3 and 12 months after the first injection based on the persistence or return of pain, with a minimum interval of 12 weeks between injections.
Arm/Group | RTX-GRT7039
All-Cause Mortality (participants affected / at risk) | 4/714
Serious Adverse Events (participants affected / at risk) | 58/714
Other Adverse Events (participants affected / at risk) | 54/714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTX-GRT7039 (N=714)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Arthritis bacterial (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Aortic valve disease (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTX-GRT7039 (N=714)
Procedural pain (Injury, poisoning and procedural complications) | 54 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT05377489/Prot_SAP_000.pdf